CLINICAL TRIAL: NCT04656457
Title: Resistance Versus Aerobic Exercises On Cancer Related Fatigue And Immunity In Breast Cancer Patients Undergoing Adjuvant Chemotherapy
Brief Title: RESISTANCE VERSUS AEROBIC EXERCISES ON Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa said tolba saleh, ASSISSTANT LECTURER, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002968
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistance exercises (Active Comparator): Resistance exercises will be involved in this technique are for upper and lower limb (Exercise program including shoulder flexion, abduction and horizontal adduction, elbow extension and flexion, calf raise, leg extension and squatting) three times daily and five times per week. The 1 repetition maximum (1RM) is measured at baseline and following the intervention. Initially, participants will do two circuits using 50% of their 1RM and repeat them 10 times for the first and second weeks, progressing to two circuits, using 60% of their 1RM and repeat 10 times for the third and fourth weeks. In fifth and sixth weeks, participants will do three circuits using 60% of their 1RM and repeat 10 times. In the last 6 weeks, patients will do three circuits using 70% of their 1RM and repeat 10 times. Time of exercise equal time of rest
  Interventions: Other: resisted exercises
- aerobic exercise (Active Comparator): Aerobic training (AT) program of submaximal intensity will include a 45-minute session five times per week under the supervision of the researcher. Aerobic exercise will consist of three phases: warm-up, training and cool down. At the beginning of exercise session, subjects will have a ten-minute warm-up. The warm up protocol will be slowly running on treadmill. Then, the warm-up phase will be followed by the training phase. At baseline, the training phase will be commenced with two 30- minute running on treadmill at 50% of their maximal heart rate (MHR) in the first week and increased to 70% MHR by the final week of training. By the end of exercise session, subjects will have a five-minute cool down. The cool down protocol will be slowly running on treadmill. The vital measures such as HR and blood pressure was monitored before patient left the department (Dimeo et al.,2016), maximum heart rate will be calculated using the formula: (HR Max =220- age)
  Interventions: Device: Treadmill

INTERVENTIONS:
Device: Treadmill — Treadmill is not used to harness power, but as exercise machines for running or walking in one place. Rather than the user powering the mill, the machine provides a moving platform with a wide conveyor belt driven by an electric motor or a flywheel. The belt moves to the rear, requiring the user to walk or run at a speed matching that of the belt. The rate at which the belt moves is the rate of walking or running. Thus, the speed of running may be controlled and measured
  Arms: aerobic exercise
Other: resisted exercises — Resistance exercises will be involved in this technique are for upper and lower limb (Exercise program including shoulder flexion, abduction and horizontal adduction, elbow extension and flexion, calf raise, leg extension and squatting)
  Arms: resistance exercises

SUMMARY:
The purpose of the study is to evaluate which is more effective resistance or aerobic exercises on cancer related fatigue and immunity in breast cancer patients undergoing adjuvant chemotherapy.

DETAILED DESCRIPTION:
The problem of cancer related fatigue and decreased immunity, as a result of treatment with adjuvant chemotherapy in breast cancer patients is not well known.

Fatigue and decreased immunity have a negative impact on work, social relationships, mood, and daily activities and cause significant impairment in overall quality of life, Furthermore the need of this study is developed from the lack of information in the published studies about the effect of the treatment with chemotherapy among breast cancer patients on inducing fatigue and decreasing immunity and the effect of resistance and aerobic exercises on improving these changes.

ELIGIBILITY:
Inclusion Criteria:

-

The subject selection will be according to the following criteria:

1. Age range from 30-60 years.
2. Females post mastectomy only will participate in the study.
3. All patients undergoing adjuvant chemotherapy and have cancer related fatigue and decreased immunity.
4. All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:

  1. Age more than 60 years or less than 30 years.
  2. Another concurrent malignant disease.
  3. Subjects suffering from any condition for which resistance or aerobic exercises contraindicated as metastasis, sever osteoporosis and cardiac diseases.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue assessment scale | The evaluation will be conducted during before the cycles
  The Fatigue Assessment Scale (FAS) is quick and easy to complete for patients, and not time consuming. It is also helpful for physicians and other health care workers in the follow-up of their patients. The FAS has proven to be a valid questionnaire to assess fatigue in cancer patients, but also in many other patients with chronic diseases
Fatigue assessment scale | The evaluation will be conducted during one and half month
  The Fatigue Assessment Scale (FAS) is quick and easy to complete for patients, and not time consuming. It is also helpful for physicians and other health care workers in the follow-up of their patients. The FAS has proven to be a valid questionnaire to assess fatigue in cancer patients, but also in many other patients with chronic diseases
Fatigue assessment scale | The evaluation will be conducted three months later
  The Fatigue Assessment Scale (FAS) is quick and easy to complete for patients, and not time consuming. It is also helpful for physicians and other health care workers in the follow-up of their patients. The FAS has proven to be a valid questionnaire to assess fatigue in cancer patients, but also in many other patients with chronic diseases
Hemoglobin level test for fatigue assessment | he evaluation will be conducted before the cycles
  Hemoglobin levels are measured by a blood test. Hemoglobin, or Hb, is usually expressed in grams per deciliter (g/dL) of blood. A low level of hemoglobin in the blood relates directly to a low level of oxygen
Hemoglobin level test for fatigue assessment | he evaluation will be conducted during one and half month
  Hemoglobin levels are measured by a blood test. Hemoglobin, or Hb, is usually expressed in grams per deciliter (g/dL) of blood. A low level of hemoglobin in the blood relates directly to a low level of oxygen
Hemoglobin level test for fatigue assessment | he evaluation will be conducted three months later
  Hemoglobin levels are measured by a blood test. Hemoglobin, or Hb, is usually expressed in grams per deciliter (g/dL) of blood. A low level of hemoglobin in the blood relates directly to a low level of oxygen
White blood cells count test for immunity assessment | he evaluation will be conducted before the cycles
  White blood cells (also called leukocytes and abbreviated as WBCs) are the cells of the immune system that are involved in protecting the body against both infectious disease and foreign invaders. All white blood cells are produced and derived from multipotent cells in the bone marrow known as hematopoietic stem cells. Leukocytes are found throughout the body, including the blood and lymphatic system
White blood cells count test for immunity assessment | he evaluation will be conducted during one and half month
  White blood cells (also called leukocytes and abbreviated as WBCs) are the cells of the immune system that are involved in protecting the body against both infectious disease and foreign invaders. All white blood cells are produced and derived from multipotent cells in the bone marrow known as hematopoietic stem cells. Leukocytes are found throughout the body, including the blood and lymphatic system
White blood cells count test for immunity assessment | he evaluation will be conducted three months later
  White blood cells (also called leukocytes and abbreviated as WBCs) are the cells of the immune system that are involved in protecting the body against both infectious disease and foreign invaders. All white blood cells are produced and derived from multipotent cells in the bone marrow known as hematopoietic stem cells. Leukocytes are found throughout the body, including the blood and lymphatic system

CONTACTS AND LOCATIONS:
Overall Officials: Amal mo abdel baky, professor, Study Director — faculty of physical therapy
Locations (1):
- Medical research institute, Alexandria, Egypt